CLINICAL TRIAL: NCT06601673
Title: Postoperative Cognitive Training for the Prevention of Delirium in Older Patients
Brief Title: Postoperative Cognitive Training to Prevent Delirium
Acronym: DELtrain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S6-2024; 2024-101267-BO-ff (Other: Ethics Committee of the Hamburg Medical Association)
Record Dates: First submitted 2024-07-30; First posted 2024-09-19 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Delirium
Keywords: older patients; frailty; neurocognitive disorder; cognitive stimulation; anaesthesia
MeSH Terms: conditions — Emergence Delirium; Frailty; Neurocognitive Disorders | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: prospective, randomized-controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention (Experimental): Tablet-based bed-side cognitive training for 2h per day for the first five days after surgery (or until discharge from hospital, if earlier).
  Interventions: Behavioral: Cognitive training
- Audio book (Sham Comparator): Listening to an audio book for 2h per day for the first five days after surgery (or until discharge from hospital, if earlier).
  Interventions: Behavioral: Listen to audio book
- Standard care (No Intervention): Standard care without any intervention.

INTERVENTIONS:
Behavioral: Cognitive training — The intervention consists of computer-based cognitive training in the areas of attention, processing speed, memory, emotional intelligence, reasoning and orientation. The training takes place under supervision for 120 minutes a day from the first to the fifth postoperative day.
  Other Names: cognitive stimulation
  Arms: Intervention
Behavioral: Listen to audio book — Here, an audio book is listened to for 2h daily for the first five postoperative days (or until discharge from hospital if earlier). The audio book is brought and set up by study staff.
  Arms: Audio book

SUMMARY:
The aim of this clinical trial is to test whether daily postoperative cognitive training can prevent delirium in older patients after major surgery.

The main questions to be answered is:

Can daily cognitive training reduce the rate of postoperative delirium in older patients after surgery?

Participants will be visited daily for the first 5 days after surgery and asked to take part in a tablet-based cognitive training programme for 2 hours a day (in 2 sessions).

The researchers will compare patients who receive the training with a control group of patients who listen to audio books for the same amount of time and a control group who receive standard care (no intervention).

DETAILED DESCRIPTION:
The most common postoperative complication in aged patients is postoperative delirium (POD), which often progresses to permanent postoperative neurocognitive disorder (pNCD). POD and pNCD are associated with significantly increased postoperative morbidity and mortality. Prevention of POD is therefore a primary therapeutic goal in the care of elderly patients. The aim of this project is to investigate the effect of cognitive stimulation on the occurrence of POD in older patients at risk after surgery.

Patients undergoing surgery who are at least 70 years old and have an increased risk of postoperative delirium will be included. The increased risk will be assessed in a preoperative assessment as part of the anaesthetic premedication consultation. It is defined as the presence of frailty (Clinical Frailty Scale, CFS and Longitudinal Urban Cohort Study Age Function Index, LUCAS-FI), cognitive impairment (Montreal Cognition Assessment Test, MoCA) or increased morbidity (Hall Risk Analysis Index). The intervention takes the form of computer-based cognitive training in the areas of attention, processing speed, memory, emotional intelligence, reasoning and orientation. Positive effects of this training have already been shown in the treatment of mild cognitive impairment (MCI), dementia and tumour-related cognitive impairment.

The training takes place under supervision for 120 minutes a day from the first to the fifth postoperative day. It is hypothesised that postoperative cognitive training can reduce the incidence of delirium in the first five days after surgery. Secondary endpoints are the reduction of neurocognitive dysfunction at one week, six weeks and six months after surgery, maintenance of function and quality of life at six months.

In order to adjust for the stimulating effects of interacting with study staff during the study visits, a control group listening to an audio book (also brought and set up by study staff) is included in the trial.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 70 years or older,
* planned surgery (abdominal surgery: general surgery, urology or gynaecology; spinal surgery, vascular medicine, cardiothoracic surgery, major trauma surgery),
* increased perioperative risk (frailty, cognitive impairment, multimorbidity).

Exclusion criteria:

* Unable to give consent,
* severe cognitive disorder or mental retardation (if training cannot be carried out)
* Insufficient knowledge of German

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium within the first five days after surgery | delirium screening twice daily from postoperative day 1-5
  Delirium screened twice daily using the 3D-Confusion Assessment Method (3D-CAM) for the first five days after surgery (0-4 hallmarks; hallmark 1+2 and 3+4 = delirium)

SECONDARY OUTCOMES:
postoperative neurocognitive disorder | postoperative day 7 (1 week after surgery)
  delayed neurocognitive recovery (compared to baseline), measured by telephone-Montreal Cognitive Assessment (MOCA) (0-15 points; 10 points or less = cognitive impairment)
postoperative neurocognitive disorder | 6 weeks after surgery
  compared to baseline, measured by telephone-MOCA (0-15 points; 10 points or less = cognitive impairment)
postoperative neurocognitive disorder | 6 months after surgery
  compared to baseline, measured by telephone-MOCA (0-15 points; 10 points or less = cognitive impairment)
Functional state (patient-reported) | 6 weeks after surgery
  compared to baseline, assessed by World Health Organization Disability Assessment (WHODAS) 2.0 questionnaire (36-item, likert scale)
Functional state (measured) | 6 weeks after surgery
  compared to baseline, assessed by functional independence measure (FIM) (18 items with 0-7 points each, less points = less functionality)
Functional state (patient-reported) | 6 months after surgery
  compared to baseline, assessed by WHODAS 2.0 questionnaire (36-item, likert scale)
Functional state (measured) | 6 months after surgery
  compared to baseline, assessed by functional independence measure (FIM) (18 items with 0-7 points each, less points = less functionality)
Quality of Life (by questionnaire) | 6 weeks after surgery
  compared to baseline, assessed by World Health Organization Quality of Life -older adults module (WHOQOL-OLD)-questionnaire (24 item, likert scale)
Quality of Life (by questionnaire) | 6 months after surgery
  compared to baseline, assessed by World Health Organization Quality of Life -older adults module (WHOQOL-OLD)-questionnaire (24 item, likert scale)
Quality of Life (by visual analogue scale) | 6 weeks after surgery
  compared to baseline, assessed by EQ-5D-5L- questionnaire (0-100 points, 100 points = best quality of life)
Quality of Life (by visual analogue scale) | 6 months after surgery
  compared to baseline, assessed by EQ-5D-5L- questionnaire (0-100 points, 100 points = best quality of life)